CLINICAL TRIAL: NCT00005168
Title: Hyperapo B and Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1042; R01HL031497 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Diabetes Mellitus; Obesity; Hypercholesterolemia, Familial
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Diabetes Mellitus; Obesity; Hyperlipoproteinemia Type II

SUMMARY:
To determine the role of apolipoprotein B and apolipoprotein A1 in the etiology of coronary artery disease.

DETAILED DESCRIPTION:
BACKGROUND:

Hyperapo B is a phenotype defined as elevated plasma level of the major apoprotein B of low density lipoproteins in the presence of a normal plasma level of low density lipoprotein cholesterol. It has been demonstrated that hyperapo B is strongly associated with coronary artery disease. In 1984 when the study began, the independence of this association with other risk factors for coronary artery disease such as cigarette smoking, hypertension, and low plasma levels of high density lipoproteins was not known. The study improved knowledge of the pathophysiology of coronary artery disease and of the genetic and biochemical defects of hyperapo B and hypoalphalipoproteinemia.

DESIGN NARRATIVE:

Interviews were conducted and clinical data collected on each index case and spouse, as well as on first degree relatives. Risk factor data included blood pressure, blood lipid levels, obesity, cigarette smoking, fasting blood sugar and diabetes, hormone use and menopause for women, physical activity, personality scores, and family history. Clinical data included the indications for coronary arteriography, history of use of lipid-lowering agents and insulin, presence of corneal arcus, xanthomata, and xanthelasma, and the electrocardiogram.

To determine if the apolipoprotein B gene and the apolipoprotein A1-C3-A4 gene cluster were independent predictors of premature coronary disease, the relation between DNA polymeric sites within the two genes and coronary disease were investigated using cloned DNA fragments as molecular probes. To determine if apolipoprotein B and apolipoprotein A levels aggregated in families and to determine if hyperapo B and hypoalphalipoproteinemia segregated as Mendelian traits, genetic analysis was conducted in the 200 index cases and the 900 first degree relatives. Studies were also conducted on the linkages between hyperapo B and haplotypes of the apolipoprotein B gene, on hyperapo B and the Ag polymorphisms, and on hyperalphalipoproteinemia and haplotypes of the apolipoprotein A1-C3-A4 gene cluster.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1984-08; Study Completion 1991-12 (Actual)

REFERENCES:
- [Background] Brunzell JD, Sniderman AD, Albers JJ, Kwiterovich PO Jr. Apoproteins B and A-I and coronary artery disease in humans. Arteriosclerosis. 1984 Mar-Apr;4(2):79-83. doi: 10.1161/01.atv.4.2.79. No abstract available. PMID 6422918
- [Background] Sniderman A, Teng B, Genest J, Cianflone K, Wacholder S, Kwiterovich P Jr. Familial aggregation and early expression of hyperapobetalipoproteinemia. Am J Cardiol. 1985 Feb 1;55(4):291-5. doi: 10.1016/0002-9149(85)90363-7. PMID 3969864
- [Background] Teng B, Sniderman A, Krauss RM, Kwiterovich PO Jr, Milne RW, Marcel YL. Modulation of apolipoprotein B antigenic determinants in human low density lipoprotein subclasses. J Biol Chem. 1985 Apr 25;260(8):5067-72. PMID 2580831
- [Background] Kwiterovich PO Jr, Bachorik PS, Franklin FA Jr, Margolis S, Georgopoulos L, Teng B, Sniderman AD. Effect of dietary treatment on the plasma levels of lipids, lipoprotein cholesterol and LDL B protein in children with type II hyperlipoproteinemia. Prog Clin Biol Res. 1985;188:123-37. PMID 4059254
- [Background] Beaty TH, Kwiterovich PO Jr, Khoury MJ, White S, Bachorik PS, Smith HH, Teng B, Sniderman A. Genetic analysis of plasma sitosterol, apoprotein B, and lipoproteins in a large Amish pedigree with sitosterolemia. Am J Hum Genet. 1986 Apr;38(4):492-504. PMID 3706300
- [Background] Genest J, Sniderman A, Cianflone K, Teng B, Wacholder S, Marcel Y, Kwiterovich P Jr. Hyperapobetalipoproteinemia. Plasma lipoprotein responses to oral fat load. Arteriosclerosis. 1986 May-Jun;6(3):297-304. doi: 10.1161/01.atv.6.3.297. PMID 3707428
- [Background] Kwiterovich P, Beaty T, Bachorik P, Chen J, Franklin F, Georgopoulos L, Sniderman A. Pediatric hyperlipoproteinemia: the phenotypic expression of hyperapobetalipoproteinemia in young probands and their parents. Prog Clin Biol Res. 1988;255:89-105. PMID 3340649
- [Background] Kwiterovich PO Jr, White S, Forte T, Bachorik PS, Smith H, Sniderman A. Hyperapobetalipoproteinemia in a kindred with familial combined hyperlipidemia and familial hypercholesterolemia. Arteriosclerosis. 1987 May-Jun;7(3):211-25. doi: 10.1161/01.atv.7.3.211. PMID 3593067
- [Background] Sniderman A, Kwiterovich PO Jr: Hyperapobetalipoproteinemia and LDL and HDL2 Heterogenity. Proceedings of the Workshop on Lipoprotein Heterogeneity, U.S. Department of Health and Human Services, NIH Publication No. 87-2646, pp 293-304, 1987
- [Background] Beaty TH, Kwiterovich PO, Laville A, Lewis B. Genetic analysis of total cholesterol and triglycerides in a pedigree of St. Thomas rabbits. J Lipid Res. 1989 Mar;30(3):387-94. PMID 2723545
- [Background] Ma YH, Ladias JA, Butler R, Schumaker VN, Antonarakis SE, Lusis AJ, Heinzman C, Kwiterovich PO. Apolipoprotein B gene haplotypes. Association between Ag and DNA polymorphisms. Arteriosclerosis. 1988 Sep-Oct;8(5):521-4. doi: 10.1161/01.atv.8.5.521. PMID 2461193
- [Background] Kwiterovich PO Jr. Biochemical, clinical, genetic and metabolic studies of hyperapo-beta-lipoproteinaemia. J Inherit Metab Dis. 1988;11 Suppl 1:57-73. doi: 10.1007/BF01800571. PMID 3141687
- [Background] Kwiterovich PO Jr. HyperapoB: a pleiotropic phenotype characterized by dense low-density lipoproteins and associated with coronary artery disease. Clin Chem. 1988;34(8B):B71-7. PMID 3042202
- [Background] Bachorik PS, Kwiterovich PO Jr. Apolipoprotein measurements in clinical biochemistry and their utility vis-a-vis conventional assays. Clin Chim Acta. 1988 Nov;178(1):1-34. doi: 10.1016/0009-8981(88)90265-3. PMID 3067911
- [Background] Ladias JA, Kwiterovich PO Jr, Smith HH, Miller M, Bachorik PS, Forte T, Lusis AJ, Antonarakis SE. Apolipoprotein B-100 Hopkins (arginine4019----tryptophan). A new apolipoprotein B-100 variant in a family with premature atherosclerosis and hyperapobetalipoproteinemia. JAMA. 1989 Oct 13;262(14):1980-8. doi: 10.1001/jama.262.14.1980. PMID 2778934
- [Background] Kwiterovich PO. Genetic influences on susceptibility to atherosclerosis in the young. Bull N Y Acad Med. 1989 Dec;65(10):1092-108; discussion 1154-60. No abstract available. PMID 2698247
- [Background] Herrington DM, Gordon GB, Achuff SC, Trejo JF, Weisman HF, Kwiterovich PO Jr, Pearson TA. Plasma dehydroepiandrosterone and dehydroepiandrosterone sulfate in patients undergoing diagnostic coronary angiography. J Am Coll Cardiol. 1990 Nov;16(6):862-70. doi: 10.1016/s0735-1097(10)80334-1. PMID 2146310
- [Background] Ladias JA, Kwiterovich PO Jr, Smith HH, Karathanasis SK, Antonarakis SE. Apolipoprotein A1 Baltimore (Arg10----Leu), a new ApoA1 variant. Hum Genet. 1990 Apr;84(5):439-45. doi: 10.1007/BF00195816. PMID 2108924
- [Background] Beaty TH, Prenger VL, Virgil DG, Lewis B, Kwiterovich PO, Bachorik PS. A genetic model for control of hypertriglyceridemia and apolipoprotein B levels in the Johns Hopkins colony of St. Thomas Hospital rabbits. Genetics. 1992 Dec;132(4):1095-104. doi: 10.1093/genetics/132.4.1095. PMID 1459430
- [Background] Prenger VL, Beaty TH, Kwiterovich PO. Genetic determination of high-density lipoprotein-cholesterol and apolipoprotein A-1 plasma levels in a family study of cardiac catheterization patients. Am J Hum Genet. 1992 Nov;51(5):1047-57. PMID 1415250
- [Background] Coresh J, Beaty TH, Kwiterovich PO Jr, Antonarakis SE. Pedigree and sib-pair linkage analysis suggest the apolipoprotein B gene is not the major gene influencing plasma apolipoprotein B levels. Am J Hum Genet. 1992 May;50(5):1038-45. PMID 1570833
- [Background] Kwiterovich PO Jr, Coresh J, Smith HH, Bachorik PS, Derby CA, Pearson TA. Comparison of the plasma levels of apolipoproteins B and A-1, and other risk factors in men and women with premature coronary artery disease. Am J Cardiol. 1992 Apr 15;69(12):1015-21. doi: 10.1016/0002-9149(92)90856-t. PMID 1561971
- [Background] Heizmann C, Kirchgessner T, Kwiterovich PO, Ladias JA, Derby C, Antonarakis SE, Lusis AJ. DNA polymorphism haplotypes of the human lipoprotein lipase gene: possible association with high density lipoprotein levels. Hum Genet. 1991 Apr;86(6):578-84. doi: 10.1007/BF00201544. PMID 1673959
- [Background] Miller M, Bell W, Plano S, Connors J, Kennedy S, Kwiterovich P. Platelet aggregation in hyperapobetalipoproteinemia. Am J Hematol. 1991 Jul;37(3):209-11. doi: 10.1002/ajh.2830370317. PMID 1858776
- [Background] Kwiterovich PO Jr, Motevalli M, Miller M, Bachorik PS, Kafonek SD, Chatterjee S, Beaty T, Virgil D. Further insights into the pathophysiology of hyperapobetalipoproteinemia: role of basic proteins I, II, III. Clin Chem. 1991 Mar;37(3):317-26. PMID 2004437
- [Background] Kwiterovich P Jr, Motevalli M, Miller M. Acylation-stimulatory activity in hyperapobetalipoproteinemic fibroblasts: enhanced cholesterol esterification with another serum basic protein, BP II. Proc Natl Acad Sci U S A. 1990 Nov;87(22):8980-4. doi: 10.1073/pnas.87.22.8980. PMID 2247473
- [Background] Miller M, Kwiterovich PO Jr. Isolated low HDL-cholesterol as an important risk factor for coronary heart disease. Eur Heart J. 1990 Dec;11 Suppl H:9-14. doi: 10.1093/eurheartj/11.suppl_h.9. PMID 2073916